CLINICAL TRIAL: NCT00942149
Title: An Open Label Study to Describe the Pharmacokinetics of Daptomycin in Infants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00019311; dapto1 (Other: DUMC)
Record Dates: First submitted 2009-07-02; First posted 2009-07-20 (Estimated); Results first posted 2012-12-12 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-06

CONDITIONS: Sepsis
Keywords: Infants; Daptomycin
MeSH Terms: conditions — Sepsis | interventions — Daptomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daptomycin cohort (Experimental)
  Interventions: Drug: Daptomycin

INTERVENTIONS:
Drug: Daptomycin — single dose of 6 mg/kg of daptomycin

SUMMARY:
This is a safety and pharmacokinetic study of single-dose daptomycin in infants > 48 hours and < 120 days of age with suspected systemic infections. The investigators will enroll a total of 24 infants in 4 gestational age/postnatal age cohorts. Interim analyses will be performed after 3 infants are enrolled in each cohort. The investigators anticipate that 6 mg/kg of daptomycin will yield an AUC <740 mch*hr/mL.

ELIGIBILITY:
Inclusion Criteria:

1. > 48 hours and <120 days of age at the time of daptomycin administration
2. Sufficient venous access to permit administration of study medication
3. Suspected to have systemic infection and appropriate cultures (blood +/- urine/CSF) are obtained within 72 hours of study entry
4. Availability and willingness of the parent/legally authorized representative to provide written informed consent

Exclusion Criteria:

1. History of anaphylaxis attributed to daptomycin
2. Previous participation in the study
3. Exposure to daptomycin in the month prior to the study
4. Serum creatinine >1.0 mg/dL
5. Concomitant administration of tobramycin

Ages: 48 Hours to 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P Brian Smith, MD MHS, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 participants were enrolled in the Duke NICU over a period of 18 months.
Groups:
- Daptomycin Cohort: There were 20 participants enrolled; each received a single 6 mg/kg dose of daptomycin IV.
Period: Overall Study
Arm/Group | Daptomycin Cohort
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Daptomycin Cohort
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 0.1 (0.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: PK of Daptomycin
Description: Area under the curve
Time Frame: 24 hours
Population: all 20 subjects were analyzed
Measure: Median (Full Range); unit: mg*h/L
Groups:
- Area Under the Curve - 24 Hours: pharmacokinetics of daptomycin
Arm/Group | Area Under the Curve - 24 Hours
Number analyzed (Participants) | 20
mg*h/L | 262.4 (.005) [166.7 to 340.2]

2. Secondary Outcome: Adverse Events Will be Monitored.
Time Frame: 7 days following last dose of study drug
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Daptomycin Cohort
Serious Adverse Events (participants affected / at risk) | 3/20
Other Adverse Events (participants affected / at risk) | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin Cohort (N=20)
Abnormal KUB (Gastrointestinal disorders) | 1 (1)
Pneumatocele (Respiratory, thoracic and mediastinal disorders) | 2 (2)
possible morgagni cdh (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daptomycin Cohort (N=20)
patent foramen ovale (Cardiac disorders) | 2 (2)
unconjugated hyperbilirubinemia (Blood and lymphatic system disorders) | 2 (2)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No